CLINICAL TRIAL: NCT04175444
Title: Establishing a Normative Database in Pediatric Population of the Head-mounted visuALL Field Analyzer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sylvia L. Groth, MD, Assistant Professor of Ophthalmology, Vanderbilt University Medical Center
Other Study IDs: 000000001
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Visual Field Defect, Peripheral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Normal Subjects: This is a study of normal subjects to establish a normative database.
  Interventions: Diagnostic Test: VisuALL Field Analyzer; Diagnostic Test: Humphrey Field Analyzer

INTERVENTIONS:
Diagnostic Test: VisuALL Field Analyzer — Each participant will conduct a visual field test with the visuaALL headset.
  Other Names: visual field testing strategy, head mounted device, Olleyes
Diagnostic Test: Humphrey Field Analyzer — Each participant will conduct a standard of care Humphrey Visual Field.
  Other Names: standard of care visual field test

SUMMARY:
The goal of this study is to determine reference values of the VisuALL Field Test in pediatric population. Standard Automatic Perimetry (SAP) is the gold standard test for the evaluation of different diseases of the visual pathway like glaucoma. Its main goal is to measure the differential light sensitivity at several locations in the central field of vision. Nevertheless, the accuracy of the current devices is limited by several factors such as the inherent inconsistency of the psychophysical test, stressful examinations and frequency of testing.

Several devices have been developed since the advent of the Octopus Perimeter and the Humphrey Field Analyzer (HFA) in an effort to improve the early detection of glaucoma. Several of these visual field test variants are implemented using laptops, iPads, and virtual reality headsets. These modalities bring portability but lack fixation methods, environmental control, and hardware standardization. These deficiencies may limit their wide usage.

The main goal of this study is to develop an initial pediatric reference database of a novel visual field test ecosystem that takes advantage of a Head Mounted Device (HMD).

DETAILED DESCRIPTION:
This is a cross-sectional observational study. The primary endpoint of the study will be at the end of the recruitment phase.

* Participants that qualify for the study will be invited to a clinical site of the Vanderbilt Eye Institute or equivalent testing space and best corrected visual acuity will be checked with standard Snellen Acuity chart.
* Once vision is confirmed to meet study requirements, the child will be instructed on how to use the headset.
* The test will be generated and participant will complete various testing strategies including suprathreshold, full threshold and individual point testing and possibly other strategies for frequency of seeing curves.
* Patient with pathology may be confirmed with formal standard of care visual field testing
* Short survey will be administered to inquire on ease of device use
* Data will be submitted for analysis

ELIGIBILITY:
Inclusion Criteria:

* No history of intraocular surgery
* Best corrected visual acuity (BVCA) 20/25 or better in each eye

Exclusion Criteria:

* A spherical refraction outside ± 5.0 D and cylinder correction outside 2.0 D.
* Intraocular surgery in the study eye
* History of systemic condition known to affect visual function.
* History of medication known to affect visual function.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population will be healthy children recruited. All ethnicities will be included and both genders.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Retinal sensitivity | End of the recruitment phase, average 3 months
  Retinal sensitivity at each location and compared between the two test strategies
Mean retinal sensitivity | End of the recruitment phase, average 3 months
  Mean retinal sensitivity at each quadrants and each hemifield

SECONDARY OUTCOMES:
Frequency of seeing curves | End of the recruitment phase, average 3 months
  Establish frequency of seeing curves with the head mounted device
Ease of device use | End of the recruitment phase, average 3 months
  Patients will be given a short survey asking about ease of device use, 2 questions on 1-5 scale with 1 being the least and 5 being the most.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Groth, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data